CLINICAL TRIAL: NCT03948750
Title: Comparison of Immunoblotting (IgA and IgG) and the Goldmann-Witmer Coefficient for Diagnosis of Ocular Toxoplasmosis in Immunocompetent Patients
Brief Title: Immunoblotting and Goldmann-Witmer Coefficient for Ocular Toxoplasmosis
Acronym: COPILOT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: COPILOT
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Ocular Toxoplasmosis
MeSH Terms: conditions — Toxoplasmosis, Ocular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Ocular Toxoplasmosis
  Interventions: Procedure: Aqueous humour sampling
- Patients without Ocular Toxoplasmosis
  Interventions: Procedure: Aqueous humour sampling

INTERVENTIONS:
Procedure: Aqueous humour sampling — Aqueous humour sampling with Goldman-Witmer coefficient and immunoblotting

SUMMARY:
Ocular toxoplasmosis (OT) is a common cause of posterior uveitis worldwide. The diagnosis of OT is based on clinical findings, but in most cases, laboratory tests are required to confirm the etiology, especially when other diseases are suspected. The aim of this study was to evaluate which methods, between the Goldmann-Witmer coefficient (GWC) and immunoblotting (IB) with both IgG and IgA, in aqueous humour (AH) samples, can be the most sensitive to diagnose OT, in current practice, especially in the first three weeks.

DETAILED DESCRIPTION:
Goldmann-Witmer coefficient (GWC): compares the levels of intraocular antibody (igG) production to that serum, as measured by ELISA.

GWC = (Level of specific IgG in aqueous humour/level of specific IgG in serum)/(Total IgG in aqueous humour/Total IgG in serum)

0.5 to 2: No intraocular antibody production, 2 to 4: Suggestive of intraocular antibody production, > 4: Diagnostic of intraocular antibody production to a specific microbial pathogen

ELIGIBILITY:
Inclusion Criteria:

* Patients who had underwent aqueous humor and serum sample for ocular toxoplasmosis diagnosis

Exclusion Criteria:

* Immunocompromised patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had underwent aqueous humor and serum sample for ocular toxoplasmosis
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-05-31 (Actual); Study Completion 2014-05-31 (Actual)

PRIMARY OUTCOMES:
Comparison of Goldmann-Witmer coefficient and immunoblotting results | Assessment of each test result at the inclusion of the patient
  All tests realized in patients were performed before their repartition in the two groups as well as the biologist could not know the status of the patient. Sensitivity and specificity were calculated for each test.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ophtalmologie, Hôpital de la Croix-Rousse (HCL), Lyon, France